CLINICAL TRIAL: NCT00168558
Title: Measles Vaccination in Guinea-Bissau. Strategies to Reduce Disease Burden and Improve Child Survival
Brief Title: Early Two-dose Measles Vaccination Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: Danish Council for Development Research (Other); Novo Nordisk A/S (Industry); AP Moeller Foundation (Other); Medical Research Council Unit, The Gambia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RUF-91134-2601-Twodose2; RUF-91134-2601; NOVO-2624; LÆGEVIDENSKABENS FREMME-2613; LÆGEVIDENSKABENS FREMME-2623
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Measles
Keywords: Non-specific effects of vaccines; Infant mortality; Child mortality; Mortality; Morbidity; Diphtheria-tetanus-pertussis vaccine; Measles vaccine; Measles; Immunisation; Low income country; Guinea-Bissau; Bandim Health Project; Immunology
MeSH Terms: conditions — Measles; Infant Death | interventions — Measles Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Standard titre Edmonston-Zagreb measles vaccine at 4½ and 9 months of age
  Interventions: Biological: Measles vaccine
- 2 (Active Comparator): Standard titre Schwarz measles vaccine at 9 months of age
  Interventions: Biological: Measles vaccine
- 3 (Active Comparator): Standard titre Edmonston-Zagreb measles vaccine at 9 months of age
  Interventions: Biological: Measles vaccine

INTERVENTIONS:
Biological: Measles vaccine — The children will be randomised to the following three arms:
  Arm 1 - Very early two-dose: V (EZ) 4½ mo of age + V (EZ) 9 mo of age.
  Arm 2 - 9 months one- or two-dose: V (SW) 9 mo of age + V (SW)/or nothing 18 mo of age.
  Arm 3 - 9 months one- or two-dose: V (EZ) 9 mo of age + V (EZ)/or nothing 18 mo of age.
  V = measles vaccination, EZ = standard titre Edmonston-Zagreb measles vaccine, SW = standard titre Schwarz measles vaccine

SUMMARY:
The specific aims are to examine in Guinea-Bissau:

* whether the standard titre Schwarz (SW) or standard-titre Edmonston-Zagreb (EZ) measles vaccine will be the best vaccine strain for use in a routine one-dose measles vaccination schedule and a two-dose measles vaccination schedule in terms of antibody response, protection against measles and child survival, and
* whether the standard-titre Edmonston-Zagreb (EZ) vaccine will be suitable for use in a very early two-dose schedule vaccinating at 4½ and 9 months of age

DETAILED DESCRIPTION:
BACKGROUND:

Two dose schedules:

After the failure of the high-titre measles vaccine, which was to be administered at 6 months of age it was suggested to perform trials of early two-dose measles vaccination schedules to lower the age of vaccination. The standard titre SW measles vaccine has been shown to be associated with a non-specific beneficial effect on child mortality that cannot be ascribed to the protection against measles. The two measles vaccines most commonly used in the Expanded Programme on Immunization (EPI) are the standard titre SW and the standard titre EZ vaccine. Surprisingly, these two vaccines have never been compared in a randomised trial with child mortality as end-point, and it is not clear which would be most suitable for use in a two-dose vaccination schedule.

From 1995 to 2002, all children in the BHP study area were included in an early two-dose measles vaccination trial from 6 months of age. The children were randomised to either a one-dose group receiving an inactivated polio vaccine (IPV) at 6 months of age and a measles vaccine at 9 months of age, or a two-dose group receiving two doses of measles vaccine at 6 and 9 months of age. For the first 6 months of the trial, the standard-titre EZ measles vaccine was used, for the rest of the trial the standard-titre SW vaccine was used. Results from the trial showed that an early two-dose schedule increased coverage considerably and provided better protection against measles among infants than the recommended one-dose at 9 months of age schedule. The EZ and the SW vaccine were used in two different cohorts - so a direct comparison was not possible, but the EZ vaccine seemed to boost a secondary immune response better than the SW vaccine. Further, the SW vaccine was less able to induce a protective level of antibodies when used from 6 months of age than the EZ vaccine. The preliminary data that we have on long-term vaccine efficacy supports that the SW vaccine might be less suitable than the EZ vaccine for use in very early measles vaccine schedules (unpublished data). On the other hand, trials performed during the 1980's in Mexico and Bangladesh have shown that administration of the standard-titre EZ vaccine to infants as young as 4-6 months of age gave good seroconversion results.

The Global Measles Strategic Plan 2001-2005 developed by the WHO and UNICEF states that all children should be guaranteed a second opportunity for measles vaccination either through campaigns or routine immunisation. The best strategy for protection of infants living in overcrowded urban African societies and who run a great risk of contracting measles before the recommended age of immunisation, will probably be early vaccination followed by a second vaccination later in childhood. If, in a vaccination campaign strategy, administration of the first vaccine is postponed this could dramatically increase the measles incidence in children below the age of vaccination. To this add that vaccination campaigns have not yet been evaluated in Africa in terms of childhood mortality relative to the routine schedule. Some children might get two, three or even more measles vaccines in an uncontrolled and not necessarily beneficial manner. Thus finding the best schedule and vaccine strain for use in a routine two-dose schedule seems a better approach for this region.

We thus propose to conduct a study comparing the standard-titre SW measles vaccine and the standard-titre EZ measles vaccine in a one- or two-dose schedule providing the first dose at 9 months of age, and then randomising the children at 18 months of age to receive either an additional dose of vaccine or nothing. The groups will be compared in terms of seroconversion-rate, proportion with an non-protective antibody level, geometric mean titer antibody level, vaccine efficacy, and child mortality. Further we plan to test the standard-titre EZ vaccine in a very early two-dose schedule providing the first dose at 4½ months of age and the second dose at 9 months of age (see also non-specific effect of vaccination).

It is likely that measles elimination vaccination campaigns will take place in the study area during the trial. The date of vaccination and the type of measles vaccine used in such campaigns will be noted, as well as simultaneous vitamin A supplementation; and the information will be included in the final data-analyses.

Non-specific effect of vaccination:

The measles vaccine has in several community studies from different parts of the world been shown to have a non-specific beneficial effect on child mortality. That means that the protection against death mediated by the vaccine exceeds the disease specific effect, ie the vaccine not only prevents deaths caused by measles, but also other deaths, presumably due to a non-specific immune stimulation providing protection from other infections than measles. For example, during the war in Guinea-Bissau that broke out on June 7, 1998, the population fled and the health care system broke down. There was no routine vaccination for at least a 3 months period. Hence, when the war started there was a group of infants who had been randomised to early SW measles vaccination at 6 months or IPV and who did not receive the standard-titre SW measles vaccine at 9 month that they would otherwise have been given. This natural experiment represents the first randomised study of the mortality effect of SW measles vaccine. The mortality ratios for measles vaccinated children were 0.29 (0.08-1.03, p=0.041) and 0.31 (0.10-0.94) over the first 3 and 7 months of the war.

Contrary to measles vaccination, diphtheria-tetanus-pertussis (DTP) vaccination has been associated with a negative effect on child mortality. Current studies indicate that the negative effect of DTP may be neutralized by a subsequent measles vaccination. The design of the proposed trial will allow us to test whether the negative effect of the DTP vaccine, which is administered by the EPI-programme at 6, 10 and 14 weeks of age, can be reverted by administration of a measles vaccine 4 weeks after the last DTP vaccination at around 4½ months of age.

Non-specific effects of vaccination are sex-specific. Girls benefit most from beneficial non-specific effects, and suffer most from apparently harmful non-specific effects of vaccination. Non-specific effects of measles vaccination may also show interaction with season, the beneficial effect of measles vaccination being largest in the dry season (unpublished), suggesting that some unknown immunological factors play a role. Season has a large influence on health in West Africa, and both morbidity and mortality, as well as immunologic parameters such as delayed-type hypersensitivity, T-cells, thymus size and measles antibody levels which are associated with season.

We intend to investigate the interactions of sex and season with measles vaccination and will assure that data on morbidity and immunologic parameters will be collected both in the dry as well as in the rainy season.

Time table:

The study began in July 2003, and with a sample size of 5.755 and a possible 2.000 children included per year, the inclusion period for the trial will be about 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Infants of 4½ months of age registered in the Bandim Health Project registration system and currently living in the Bandim Health Project areas: Bandim I, Bandim II, Belem, Mindará and Cuntum; and who received all three diphtheria-tetanus-pertussis vaccinations at least 4 weeks before enrollment

Exclusion Criteria:

* Severe illness requiring immediate hospitalisation

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5879 (Actual)
Dates: Start 2003-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Vaccine efficacy | Assessed by study completion
Measles specific mortality | Assessed by study completion
All cause sex-specific mortality until 3 years of age | Assessed by study completion

SECONDARY OUTCOMES:
Measles antibody level at 4½, 9, 18 and 24 months of age | Assessed by study completion
Morbidity from 4½ to 12 months of age | Assessed by study completion
Anthropometric measures at 4½, 9, 18 and 24 months of age | Assessed by study completion

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, MSc, Dr. Med, Study Director — Bandim Health Project; May-Lill Garly, PHD, DTM&H, Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Bissau, Apartado 861, Guinea-Bissau

REFERENCES:
- [Derived] Brond M, Martins CL, Byberg S, Benn CS, Whittle H, Garly ML, Aaby P, Fisker AB. Randomized Trial of 2 Versus 1 Dose of Measles Vaccine: Effect on Hospital Admission of Children After 9 Months of Age. J Pediatric Infect Dis Soc. 2018 Aug 17;7(3):226-233. doi: 10.1093/jpids/pix042. PMID 28992261
- [Derived] Rasmussen SM, Biering-Sorensen S, Byberg S, Andersen A, Bjerregaard-Andersen M, Rodrigues A, Benn CS, Martins CL, Aaby P. The effect of early measles vaccination at 4.5 months of age on growth at 9 and 24 months of age in a randomized trial in Guinea-Bissau. BMC Pediatr. 2016 Dec 3;16(1):199. doi: 10.1186/s12887-016-0738-z. PMID 27912735
- [Derived] Benn CS, Martins CL, Fisker AB, Diness BR, Garly ML, Balde I, Rodrigues A, Whittle H, Aaby P. Interaction between neonatal vitamin A supplementation and timing of measles vaccination: a retrospective analysis of three randomized trials from Guinea-Bissau. Vaccine. 2014 Sep 22;32(42):5468-74. doi: 10.1016/j.vaccine.2014.07.090. Epub 2014 Aug 13. PMID 25131735
- [Derived] Aaby P, Martins CL, Garly ML, Andersen A, Fisker AB, Claesson MH, Ravn H, Rodrigues A, Whittle HC, Benn CS. Measles vaccination in the presence or absence of maternal measles antibody: impact on child survival. Clin Infect Dis. 2014 Aug 15;59(4):484-92. doi: 10.1093/cid/ciu354. Epub 2014 May 14. PMID 24829213
- [Derived] Martins C, Garly ML, Bale C, Rodrigues A, Njie-Jobe J, Benn CS, Whittle H, Aaby P. Measles virus antibody responses in children randomly assigned to receive standard-titer edmonston-zagreb measles vaccine at 4.5 and 9 months of age, 9 months of age, or 9 and 18 months of age. J Infect Dis. 2014 Sep 1;210(5):693-700. doi: 10.1093/infdis/jiu117. Epub 2014 Mar 31. PMID 24688075
- [Derived] Martins CL, Benn CS, Andersen A, Bale C, Schaltz-Buchholzer F, Do VA, Rodrigues A, Aaby P, Ravn H, Whittle H, Garly ML. A randomized trial of a standard dose of Edmonston-Zagreb measles vaccine given at 4.5 months of age: effect on total hospital admissions. J Infect Dis. 2014 Jun 1;209(11):1731-8. doi: 10.1093/infdis/jit804. Epub 2014 Jan 16. PMID 24436454
- [Derived] Martins C, Garly ML, Bale C, Rodrigues A, Benn CS, Whittle H, Aaby P. Measles antibody levels after vaccination with Edmonston-Zagreb and Schwarz measles vaccine at 9 months or at 9 and 18 months of age: a serological study within a randomised trial of different measles vaccines. Vaccine. 2013 Nov 19;31(48):5766-71. doi: 10.1016/j.vaccine.2013.08.044. Epub 2013 Aug 28. PMID 23994379
- [Derived] Aaby P, Martins CL, Garly ML, Bale C, Andersen A, Rodrigues A, Ravn H, Lisse IM, Benn CS, Whittle HC. Non-specific effects of standard measles vaccine at 4.5 and 9 months of age on childhood mortality: randomised controlled trial. BMJ. 2010 Nov 30;341:c6495. doi: 10.1136/bmj.c6495. PMID 21118875
- [Derived] Martins CL, Garly ML, Bale C, Rodrigues A, Ravn H, Whittle HC, Lisse IM, Aaby P. Protective efficacy of standard Edmonston-Zagreb measles vaccination in infants aged 4.5 months: interim analysis of a randomised clinical trial. BMJ. 2008 Jul 24;337:a661. doi: 10.1136/bmj.a661. PMID 18653640
- See also: Statens Serum Institut, Denmark — http://www.ssi.dk